CLINICAL TRIAL: NCT04080739
Title: Regional Block for Postoperative Free Flap Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Anthony Morlandt, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003574
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): US-guided ipsilateral sciatic nerve block for fibula free flap patients utilizing ropivacaine 0.2% at 2-8 cc/hr for fibula free flap patients; US-guided infraclavicular brachial plexus nerve block for forearm free lap patients utilizing ropivacaine 0.2% at 2-8cc/hr for forearm free flap patients.
  Interventions: Drug: ropivicaine 0.2%
- Control Group (No Intervention): No regional anesthetic of any kind during the surgical procedure.

INTERVENTIONS:
Drug: ropivicaine 0.2% — 2-8 cc/hr of 0.2% ropivicaine given as a regional block via US-guided ipsilateral sciatic nerve block for fibula free flap patients or US-guided infraclavicular brachial plexus nerve block for forearm free flap patients.
  Other Names: Naropin
  Arms: Experimental Group

SUMMARY:
The purpose of this protocol is to evaluate the safety and efficacy of regional anesthesia for head and neck patients undergoing microvascular free flap reconstruction.

DETAILED DESCRIPTION:
The increasing rate of opioid related overdose mortality is well documented in the literature and approached 15 per 100,000 in 2017. Because of a growing epidemic in the US, the medical community is under scrutiny to curtail opioid prescription. However, this is weighed against surgical outcomes; importantly, postoperative pain has adverse effects on function, recovery and quality of life.

Regional anesthesia provides a non opioid based, pain control strategy. First, regional anesthesia decreases systemic adverse events including respiratory failure in abdominal surgery, decreases length of stay and improves rehabilitation in common orthopedic procedures such as total knee arthroplasty and shoulder arthroplasty. Second, the physiologic benefits of regional anesthesia are compelling including augmented micro and macrocirculation, maintenance of body temperature and decreased systemic stress response through chemical sympathectomy. Finally, regional anesthesia has been established as safe in the microvascular and anesthesia literature for pediatric, and adult patients.

ELIGIBILITY:
Inclusion criteria:

* Age > 18
* Able to consent for themselves
* Undergoing a head and neck surgery at UAB with reconstruction using either a forearm free flap or a fibula free flap

Exclusion criteria:

* Age < 18
* Unable to consent for themselves
* Non-English speakers
* Non-resectable tumor
* Have a known opioid tolerance, or are on a home opioid regimen for a chronic condition. (Short-term opioid use for diagnostic procedures (i.e. biopsy) or new cancer diagnosis will be allowed).
* Patients with known hepatic failure, renal failure, or sulfa allergy, as determined by standard of care labs drawn within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Morlandt, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Le JM, Gigliotti J, Sayre KS, Morlandt AB, Ying YP. Supplemental Regional Block Anesthesia Reduces Opioid Utilization Following Free Flap Reconstruction of the Oral Cavity: A Prospective, Randomized Clinical Trial. J Oral Maxillofac Surg. 2023 Feb;81(2):140-149. doi: 10.1016/j.joms.2022.10.015. Epub 2022 Nov 1. PMID 36442533
- See also: Journal of Oral and Maxillofacial Surgery, Published November 1, 2022 — https://doi.org/10.1016/j.joms.2022.10.015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 50 | 50
Completed | 48 | 50
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 44 | 47 | 91
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 56 [16 to 81] | 56 [16 to 81] | 56 [16 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Opioid Utilization Measured in Oral Morphine Equivalent (OME)
Description: Opioid Utilization was measured by the number of mg of Oral Morphine Equivalent (oral pain medication) was given to patients.
Time Frame: 21 days
Population: Subjects included
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
mg | 118 [19.81 to 217.05] | 166 [35.66 to 296.98]

2. Secondary Outcome: Opioid Medication Use
Description: Amount of opioid medication used post-operatively
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: morphine milliequivalents
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
morphine milliequivalents | 118 (98.6) | 166 (130.7)

ADVERSE EVENTS:
Time Frame: 5 days post procedure
Description: No adverse events were reported.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT04080739/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT04080739/ICF_001.pdf